CLINICAL TRIAL: NCT03701490
Title: A Proof of Concept, Randomized, Controlled Clinical Trial to Assess the Efficacy of Subcutaneous Progesterone (Prolutex) Versus Vaginal Progesterone (Progeffik) for Endometrial Preparation in Women Undergoing Frozen Embryo Transfer(FET) Cycles
Brief Title: Prolutex in Frozen Embryo Transfer Cycles At the Blastocyst Stage (PROGEX)
Acronym: PROGEX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IBSA Institut Biochimique SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18E-Prg06
Record Dates: First submitted 2018-10-08; First posted 2018-10-10 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2023-02

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prolutex (Experimental)
  Interventions: Drug: Progesterone subcutaneous
- Progeffik (Experimental)
  Interventions: Drug: Progesterone Vaginal Product

INTERVENTIONS:
Drug: Progesterone subcutaneous — 25 mg/twice a day.
  Arms: Prolutex
Drug: Progesterone Vaginal Product — 200 mg three times a day.
  Arms: Progeffik

SUMMARY:
The objective of this proof of concept clinical trial is to evaluate the impact of two different progesterone treatments for endometrial preparation (25 mg/twice-a-day, subcutaneous injection, and 200 mg/three times a day, vaginal administration) on the clinical pregnancy rate in women undergoing frozen embryo transfer (FET) at blastocyst stage.

ELIGIBILITY:
Inclusion Criteria:

* Women attending the clinics to undergo a frozen blastocyst embryo transfer, having given written informed consent, with the following characteristics:
* 18-49 years of age for subjects undergoing ET with donated oocytes (both inclusive);
* 18-37 years of age for subjects undergoing ET with autologous oocytes (both inclusive);
* BMI <32 kg/m2;
* Adequate endometrium preparation (Endometrial thickness > 7 mm) and E2 levels ( >100 pg/ml) on the day progesterone treatment is started;
* P4 levels <1.5 ng/ml on the day progesterone treatment is started;
* Transfer of 1 or 2 frozen embryos at blastocyst stage
* Transfer of frozen embryos of quality A and/or B according to Gardner criteria1;
* Semen from ejaculation either from the partner or from a bank
* ≤ 3 previous ET (frozen and fresh) with no pregnancy
* Normal uterine cavity (i.e. no polyp or protruding sub-mucosal fibroid).

Exclusion Criteria:

* Presence of functional follicles > 10 mm of diameter on the day progesterone treatment is started;
* Intramural uterine fibroids that distort the uterine cavity or polyps >1 cm;
* Stage III or IV endometriosis (endometriomas);
* Hydrosalpinx;
* Pregnancy or lactation
* Malformations of the sexual organs incompatible with pregnancy;
* Patients affected by pathologies associated with any contraindication of being pregnant;
* Known allergy to progesterone preparations or their excipients;
* Uncontrolled adrenal or thyroid dysfunction;
* Undiagnosed vaginal haemorrhage;
* History of, or current arterial disease;
* Patients with hepatic impairment;
* HIV, Hepatitis B Virus or Hepatitis C Virus seropositive;
* Neoplasias (current) or history of neoplasia that may be responsive to progesterone;
* High grade cervical dysplasia;
* Active thrombophlebitis or thromboembolic disorders, or a history of hormone-associated thrombophlebitis or thromboembolic disorders;
* Currently dependent on alcohol, drugs or psychotropic drugs
* History of recurrent pregnancy loss defined as 3 or more spontaneous miscarriages wherein pregnancy developed to a minimum of a gestational sac on transvaginal ultrasonography;
* Participation in a concurrent clinical trial or another trial within the past 2 months;
* Use of concomitant medications that might interfere with the study evaluation: hormonal treatments other than those used in the study, except thyroid hormones.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 213 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2022-09-28 (Actual); Study Completion 2022-12-03 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 4-5 weeks after progesterone treatment start.

SECONDARY OUTCOMES:
Serum progesterone level | 19+/-2 days and 4-5 weeks after start progesterone treatment
Frequency of uterine contractions | on the day of Embryo transfer (i.e. 5 days after start progesterone treatment)
  n of uterine contraction/min
Positive serum pregnancy (beta-hCG) test rate | 19+/-2 days after start progesterone treatment
Implantation rate | 4-5 weeks after start progesterone treatment.
Ongoing pregnancy rate | 9-11 weeks after start progesterone treatment.
Abortion rate | 9 months after start progesterone treatment.

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Instituto Bernabeu, Alicante
  - Instituto Bernabeu Madrid, Madrid
  - Ginemed, Seville

IPD SHARING:
Plan to Share IPD: No